CLINICAL TRIAL: NCT05035212
Title: A PHASE 3 STUDY TO EVALUATE THE EFFICACY, IMMUNOGENICITY, AND SAFETY OF RESPIRATORY SYNCYTIAL VIRUS (RSV) PREFUSION F SUBUNIT VACCINE IN ADULTS
Brief Title: Study to Evaluate the Efficacy, Immunogenicity, and Safety of RSVpreF in Adults.
Acronym: RENOIR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C3671013; 2021-003693-31 (EudraCT Number)
Record Dates: First submitted 2021-08-20; First posted 2021-09-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Lower Respiratory Tract Illness
Keywords: Lower Respiratory Tract Illness; RSV; Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Efficacy Study: RSVpreF vaccine (Experimental): RSVpreF
  Interventions: Biological: RSVpreF
- Efficacy Study: Placebo dose (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- SSA: Vaccination of RSVpreF recipients with RSVpreF (Year 2 revaccination) (Experimental): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSA will receive RSVpreF in SSA.
  Interventions: Biological: RSVpreF
- SSA: Vaccination of RSVpreF recipients with Placebo (Placebo Comparator): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSA will receive Placebo in SSA.
  Interventions: Biological: Placebo
- SSB: Vaccination of RSVpreF recipients with RSVpreF (Year 1 revaccination) (Experimental): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSB will receive RSVpreF in SSB.
  Interventions: Biological: RSVpreF
- SSB: Vaccination of RSVpreF recipients with Placebo (Placebo Comparator): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSB will receive Placebo in SSB.
  Interventions: Biological: Placebo
- SSC: Vaccination of RSVpreF recipients with RSVpreF (Year 3 revaccination) (Experimental): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSC will receive RSVpreF at the Year 3 vaccination followed by placebo at the Year 4 vaccination in SSC.
  Interventions: Biological: RSVpreF
- SSC: Vaccination of RSVpreF recipients with RSVpreF (Year 4 revaccination) (Experimental): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSC will receive placebo at the Year 3 vaccination followed by RSVpreF at the Year 4 vaccination in SSC.
  Interventions: Biological: RSVpreF
- SSC: Vaccination of RSVpreF recipients with Placebo (Placebo Comparator): Participants who originally received RSVpreF in the Efficacy Study and are eligible for SSC will receive placebo at both the Year 3 and Year 4 vaccination in SSC.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVpreF — RSV vaccine (RSVpreF)
  Arms: Efficacy Study: RSVpreF vaccine; SSA: Vaccination of RSVpreF recipients with RSVpreF (Year 2 revaccination); SSB: Vaccination of RSVpreF recipients with RSVpreF (Year 1 revaccination); SSC: Vaccination of RSVpreF recipients with RSVpreF (Year 3 revaccination); SSC: Vaccination of RSVpreF recipients with RSVpreF (Year 4 revaccination)
Biological: Placebo — Placebo
  Arms: Efficacy Study: Placebo dose; SSA: Vaccination of RSVpreF recipients with Placebo; SSB: Vaccination of RSVpreF recipients with Placebo; SSC: Vaccination of RSVpreF recipients with Placebo

SUMMARY:
Efficacy Study: This randomized, double-blinded, placebo-controlled Phase 3 study is designed to assess the safety, immunogenicity, and efficacy of a single dose of RSVpreF in the prevention of LRTI-RSV in adults:

* At a dose of 120µg.
* In adults 60 years of age and older.
* The duration of the study for each participant will be up to approximately 24 months.
* The study will be conducted in the United States, Canada, Netherlands, Finland, Argentina, Japan and South Africa.

Substudy A: This study is an extension of the efficacy study and was designed to evaluate the safety and immunogenicity of a second dose of RSVpreF when administered after a dosing interval of approximately 2 years:

* At a dose of 120µg (as studied in the Phase 3 Efficacy Study)
* Blood samples will be collected for antibody testing.
* The duration of the study for each participant will be up to approximately 18 months.
* The study will be conducted in the United States and Argentina.

Substudy B: This study was designed to evaluate the safety and immunogenicity of a second dose of RSVpreF when administered after a dosing interval of approximately 1 year:

* At a dose of 120µg (as studied in the Phase 3 Efficacy Study)
* Blood samples will be collected for antibody testing.
* The duration of the study for each participant will be up to approximately 18 months.
* The study will be conducted in Argentina.

Substudy C: This study was designed to evaluate the safety and immunogenicity of a second dose of RSVpreF when administered after a dosing interval of either 3 or 4 years:

* At a dose of 120µg (as studied in the Phase 3 Efficacy Study)
* Participants will receive either placebo or a second dose of RSVpreF approximately 3 or 4 years after receiving the initial dose of RSVpreF in the main efficacy study.
* Blood samples will be collected for antibody testing.
* The duration of the study for each participant will be up to approximately 24 months.
* The study will be conducted in the United States and Canada.

ELIGIBILITY:
Efficacy Study

Inclusion Criteria:

* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, frequent symptom assessment by mobile device application, and other study procedures, including collection of nasal swabs by themselves and by study staff when indicated.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for participants with known stable infection with HIV, HCV, or HBV can be found in the protocol.

* Adults who are ambulatory and live in the community, or in assisted living or long-term care residential facilities that provide minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
* Male or female participants ≥60 years of age.

  * Male participants able to father children must agree to use a highly effective method of contraception from the time of informed consent through at least 28 days after study intervention administration.
  * Female participants must not be of childbearing potential.

Exclusion Criteria:

* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
* Serious chronic disorder including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-months follow-up visit (Visit 3).

Note: This criterion does not apply to participants who are participating in a follow-up period for another study involving a study intervention that is an investigational drug or vaccine, if receipt of the last dose was at least 6 months prior to consenting for this study and there is no further dosing anticipated from the previous study during the participant's participation in this study - Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

Note: Participants with COPD or asthma can be enrolled if chronic corticosteroids do not exceed a dose equivalent to 10 mg/day of prednisone.

* Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Substudy A

Inclusion Criteria:

* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, frequent symptom assessment by mobile device application, and other study procedures, including collection of nasal swabs by themselves and by study staff when indicated.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for participants with known stable infection with HIV, HCV, or HBV can be found in the protocol.

* Adults who are ambulatory and live in the community, or in assisted living or long-term care residential facilities that provide minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
* Male or female participants ≥60 years of age.

  * Male participants able to father children must agree to use a highly effective method of contraception from the time of informed consent through at least 28 days after study intervention administration.
  * Female participants must not be of childbearing potential.
* Participants who received RSVpreF in the efficacy study.
* Participants who have a Visit 2 serology sample available for testing from the efficacy study, completed the end-of-Season 2 visit (Visit 5), and did not meet exclusion criteria throughout the efficacy study duration.

Exclusion Criteria:

* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
* Serious chronic disorder including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-months follow-up visit (Visit 103).

Note: This criterion does not apply to participants who are participating in a follow-up period for another study involving a study intervention that is an investigational drug or vaccine, if receipt of the last dose was at least 6 months prior to consenting for this study and there is no further dosing anticipated from the previous study during the participant's participation in this study

- Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

Note: Participants with COPD or asthma can be enrolled if chronic corticosteroids do not exceed a dose equivalent to 10 mg/day of prednisone.

* Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.

Note: This criterion does not include the receipt of RSVpreF in the efficacy study. Per inclusion criterion #6, receipt of RSVpreF in the efficacy study is required to participate in Substudy A.

* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participant was confirmed by the sponsor to have previously received the study intervention more than once.

Substudy B

Inclusion Criteria:

* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, frequent symptom assessment by mobile device application, and other study procedures, including collection of nasal swabs by themselves and by study staff when indicated.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for participants with known stable infection with HIV, HCV, or HBV can be found in the protocol.

* Adults who are ambulatory and live in the community, or in assisted living or long-term care residential facilities that provide minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
* Male or female participants ≥60 years of age.

  * Male participants able to father children must agree to use a highly effective method of contraception from the time of informed consent through at least 28 days after study intervention administration.
  * Female participants must not be of childbearing potential. 6. Participants who received RSVpreF in the efficacy study.
* Participants who received RSVpreF in the efficacy study.
* Participants who have a Visit 2 serology sample available for testing from the efficacy study and did not meet exclusion criteria through Visit 4 of the efficacy study.

Exclusion Criteria:

* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
* Serious chronic disorder including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-months follow-up visit (Visit 203).

Note: This criterion does not apply to participants who are participating in a follow-up period for another study involving a study intervention that is an investigational drug or vaccine, if receipt of the last dose was at least 6 months prior to consenting for this study and there is no further dosing anticipated from the previous study during the participant's participation in this study - Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

Note: Participants with COPD or asthma can be enrolled if chronic corticosteroids do not exceed a dose equivalent to 10 mg/day of prednisone.

* Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.

Note: This criterion does not include the receipt of RSVpreF in the efficacy study. Per inclusion criterion #6, receipt of RSVpreF in the efficacy study is required to participate in Substudy B.

* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participant was confirmed by the sponsor to have previously received the study intervention more than once.
* Participants who completed Vaccination 1 from the efficacy study less than 9 months or greater than 15 months prior to revaccination.

Substudy C

Inclusion Criteria:

* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, frequent symptom assessment by mobile device application, and other study procedures, when indicated.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for participants with known stable infection with HIV, HCV, or HBV can be found in the protocol.

* Adults who are ambulatory and live in the community, or in assisted living or long-term care residential facilities that provide minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
* Male or female participants ≥60 years of age.
* Participants who received RSVpreF in the efficacy study.
* Participants who have a Visit 2 serology sample available for testing from the efficacy study, completed the end-of-Season 2 visit (Visit 5), and did not meet exclusion criteria throughout the efficacy study duration.

Exclusion Criteria:

* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s) or any related vaccine.
* Serious chronic disorder including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participation in other studies involving an investigational product within 28 days prior to consent and/or through and including the 6-months follow-up visit (Visit 303 or Visit 306).

Note: This criterion does not apply to participants who are participating in a follow-up period for another study involving a study intervention that is an investigational drug or vaccine, if receipt of the last dose was at least 6 months prior to consenting for this study and there is no further dosing anticipated from the previous study during the participant's participation in this study

- Individuals who receive chronic systemic treatment with immunosuppressive therapy, including cytotoxic agents, monoclonal antibodies, systemic corticosteroids, or radiotherapy, eg, for cancer or an autoimmune disease, from 60 days before study intervention administration or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

Note: Participants with COPD or asthma can be enrolled if chronic corticosteroids do not exceed a dose equivalent to 10 mg/day of prednisone.

* Receipt of blood/plasma products or immunoglobulin within 60 days before study intervention administration.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.

Note: This criterion does not include the receipt of RSVpreF in the efficacy study. Per inclusion criterion #6, receipt of RSVpreF in the efficacy study is required to participate in Substudy C.

* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participant was confirmed by the sponsor to have previously received the study intervention more than once.
* Prior history of any subtype of Guillain-Barré syndrome of any etiology.
* Current or prior participation in Substudy A or Substudy B.
* Participants who completed Vaccination 1 from the efficacy study less than 32 months or greater than 40 months prior to revaccination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38861 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Efficacy Study: Number of first episode of RSV-associated lower respiratory tract illness (LRTI-RSV) in the first RSV season | From Day 15 after vaccination until the end of season 1 visit (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 2 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 3 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Proportion of participants reporting prompted local reactions within 7-days after vaccination | Within 7 days after vaccination
  Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity
Efficacy Study: Proportion of participants reporting prompted systemic events within 7-days after vaccination | Within 7 days after vaccination
  Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
Efficacy Study: Proportion of participants reporting AE within 1-month after vaccination | Within 1 month after vaccination (up to 35 days)
  An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
Efficacy Study: Proportion of participants reporting SAE throughout the study | Throughout the study duration (an average of 30 months)
  SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Efficacy Study: Proportion of participants reporting NDCMC throughout the study | Throughout the study duration (an average of 30 months)
  An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects (eg, asthma).
SSA: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 2-dose of RSVpreF | Before revaccination and 1, 6, 12 and 18-months after revaccination with RSVpreF in SSA
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs), and geometric mean fold rise (GMFR). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSA: Proportion of participants reporting prompted local reactions within 7-days after revaccination | Within 7 days after revaccination
  Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity
SSA: Proportion of participants reporting prompted systemic events within 7-days after revaccination | Within 7 days after revaccination
  Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
SSA: Proportion of participants reporting AE within 1-month after revaccination | Within 1 month after revaccination (up to 35 days)
  An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
SSA: Proportion of participants reporting SAE throughout the study | Throughout the study duration (approximately 18 months)
  SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
SSA: Proportion of participants reporting NDCMC throughout the study | Throughout the study duration (approximately 18 months)
  An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects (eg, asthma).
SSB: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 2-dose of RSVpreF | Before revaccination and 1, 6, 12 and 18-months after revaccination with RSVpreF in SSB
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs), and geometric mean fold rise (GMFR). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSB: Proportion of participants reporting prompted local reactions within 7-days after revaccination | Within 7 days after revaccination
  Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity.
SSB: Proportion of participants reporting prompted systemic events within 7-days after revaccination | SSB: Proportion of participants reporting prompted systemic events within 7-days after revaccination
  Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
SSB: Proportion of participants reporting AE within 1-month after revaccination | Within 1 month after revaccination (up to 35 days)
  An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
SSB: Proportion of participants reporting SAE throughout the study | Throughout the study duration (approximately 18 months)
  SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
SSB: Proportion of participants reporting NDCMC throughout the study | Throughout the study duration (approximately 18 months)
  An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects (eg, asthma).
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received RSVpreF or placebo in SSC (Year 3) | 1 month after revaccination in SSC (Year 3)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean NT ratios. The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 1 dose in the Main Efficacy Study (preS2) and revaccination in SSC (Year 3) | At preseason 2 (preS2) after receiving the initial vaccination in the efficacy study and 1 month after revaccination in SSC (Year 3)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean NT ratios. The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 1 dose in the Main Efficacy Study and revaccination in SSC (Year 3) | 1 month after receiving the initial vaccination in the efficacy study and 1 month after revaccination in SSC (Year 3)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean of individual NT ratios (GMIR). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received RSVpreF or placebo in SSC (Year 4) | 1 month after revaccination in SSC (Year 4)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean NT ratios. The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 1 dose in the Main Efficacy Study (preS2) and revaccination in SSC (Year 4) | At preseason 2 (preS2) after receiving the initial vaccination in the efficacy study and 1 month after revaccination in SSC (Year 4)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean NT ratios. The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received 1 dose in the Main Efficacy Study and revaccination in SSC (Year 4) | 1 month after receiving the initial vaccination in the efficacy study and 1 month after revaccination in SSC (Year 4)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean of individual NT ratios (GMIR). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Proportion of participants reporting prompted local reactions within 7-days after revaccination (Year 3) | Within 7 days after revaccination
  Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity.
SSC: Proportion of participants reporting prompted local reactions within 7-days after revaccination (Year 4) | Within 7 days after revaccination
  Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity.
SSC: Proportion of participants reporting prompted systemic events within 7-days after revaccination (Year 3) | Within 7 days after revaccination
  Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
SSC: Proportion of participants reporting prompted systemic events within 7-days after revaccination (Year 4) | Within 7 days after revaccination
  Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
SSC: Proportion of participants reporting AE within 1-month after revaccination (Year 3) | Within 1 month after revaccination (up to 35 days)
  An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
SSC: Proportion of participants reporting AE within 1-month after revaccination (Year 4) | Within 1 month after revaccination (up to 35 days)
  An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
SSC: Proportion of participants reporting SAE after revaccination (Year 3) | Following revaccination and throughout the study duration (approximately 24 months)
  SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
SSC: Proportion of participants reporting SAE after revaccination (Year 4) | Following revaccination and throughout the study duration (approximately 12 months)
  SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
SSC: Proportion of participants reporting NDCMC after revaccination (Year 3) | Following revaccination and throughout the study duration (approximately 24 months)
  An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects (eg, asthma).
SSC: Proportion of participants reporting NDCMC after revaccination (Year 4) | Following revaccination and throughout the study duration (approximately 12 months)
  An NDCMC is defined as a disease or medical condition, not previously identified, that is expected to be persistent or otherwise long-lasting in its effects (eg, asthma).

SECONDARY OUTCOMES:
Efficacy Study: Number of first episode of RSV-associated severe LRTI (sLRTI-RSV) in the first RSV season | From Day 15 after vaccination until the end of season 1 visit (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. sLRTI-RSV is defined as LRTI-RSV with at least 1 of the conditions: 1)Hospitalization due to LRTI-RSV; 2)New/increased oxygen supplementation; 3)New/increased mechanical ventilation
Efficacy Study: Number of first episode of LRTI-RSV in the second RSV season | During the second RSV season (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 2 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 3 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Number of first episode of LRTI-RSV across 2 RSV seasons | From Day 15 after vaccination until the end of season 2 visit (an average of 12 months of surveillance)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 2 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. LRTI-RSV is defined as an ARI with 3 or more of the lower respiratory signs/symptoms lasting more than 1 day during the same illness, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Number of first episode of RSV-associated ARI (ARI-RSV) in the first RSV season | From Day 15 after vaccination until the end of season 1 visit (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. ARI-RSV is defined as an ARI with at least 1 signs/symptoms lasting more than 1 day, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Number of first episode of ARI-RSV in the second RSV season | During the second RSV season (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. ARI-RSV is defined as an ARI with at least 1 signs/symptoms lasting more than 1 day, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Number of first episode of ARI-RSV across 2 RSV seasons | From Day 15 after vaccination until the end of season 2 visit (an average of 12 months of surveillance)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. ARI-RSV is defined as an ARI with at least 1 signs/symptoms lasting more than 1 day, plus RT-PCR-confirmed RSV infection within 7 days of ARI symptom onset.
Efficacy Study: Number of first episode of sLRTI-RSV in the second RSV season | During the second RSV season (an average of 6 months)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. sLRTI-RSV is defined as LRTI-RSV with at least 1 of the conditions: 1)Hospitalization due to LRTI-RSV; 2)New/increased oxygen supplementation; 3)New/increased mechanical ventilation
Efficacy Study: Number of first episode of sLRTI-RSV across 2 RSV seasons | From Day 15 after vaccination until the end of season 2 visit (an average of 12 months of surveillance)
  Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR)-confirmed RSV A and/or RSV B- associated acute respiratory illness (ARI) is assessed. sLRTI-RSV is defined as LRTI-RSV with at least 1 of the conditions: 1)Hospitalization due to LRTI-RSV; 2)New/increased oxygen supplementation; 3)New/increased mechanical ventilation
Efficacy Study: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers | Before vaccination, 1-month after vaccination, before season 2 (approximately 12 months after vaccination)
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs), and geometric mean fold rise (GMFR). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSA: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received placebo in SSA. | Before revaccination and 1, 6, 12 and 18-months after revaccination with placebo in SSA
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSB: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received placebo in SSB | Before revaccination and 1, 6, 12 and 18-months after revaccination with placebo in SSB
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.
SSC: Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B neutralizing titers from participants who received placebo in SSC. | Participants receiving placebo at the Year 3 vaccination: 1 month, 3 and 3.5 years after efficacy study vaccination
  RSV A and RSV B neutralizing titers (NT), expressed as Geometric Mean Titers (GMTs). The NTs were calculated as the interpolated reciprocal of the serum dilution resulting in 50% reduction in the number of viral focus forming units when compared to the control without test serum.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (259):
- United States (173):
  - St. Vincent's Birmingham (Pharmacy), Birmingham, Alabama
  - St. Vincent's Birmingham, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Lenzmeier Family Medicine / Avacare, Glendale, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Cognitive Clinical Trials, LLC, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - HOPE Research Institute, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - The Institute for Liver Health dba Arizona Clinical Trials, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - eStudySite, Chula Vista, California
  - Benchmark Research, Colton, California
  - West Coast Research, Dublin, California
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - Chemidox Clinical Trials, Lancaster, California
  - Ark Clinical Research, Long Beach, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Clinica mi Salud by Focil Med, Oxnard, California
  - De Silva Medical Inc, Palmdale, California
  - Empire Clinical Research, Pomona, California
  - Paradigm Clinical Research Center, Redding, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Benchmark Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Tekton Research LLC, Longmont, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - IDEAL Clinical Research, Aventura, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - Invictus Clinical Research Group, LLC, Coconut Creek, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Universal Axon Clinical Research, LLC (Administrative), Doral, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Doral Medical Research, LLC, Hialeah, Florida
  - M3 Wake Research - Lake City, Lake City, Florida
  - Optimus U Corporation, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - De La Cruz Research Center, LLC, Miami, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - IDEAL Clinical Research, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Headlands Research Sarasota, Sarasota, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Conquest Research, Winter Park, Florida
  - Javara - Privia Medical Group Georgia - Albany, Albany, Georgia
  - Coastal Heritage Clinical Research, Hinesville, Georgia
  - Javara - Privia Medical Group Georgia - Savannah, Savannah, Georgia
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Javara Inc., Thomasville, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Great Lakes Clinical Trials, LLC dba Flourish Research, Chicago, Illinois
  - DM Clinical Research, Melrose Park, Illinois
  - Affinity Health Corp, Oak Brook, Illinois
  - Accellacare - DuPage, Oak Lawn, Illinois
  - MOC Research, Mishawaka, Indiana
  - Velocity Clinical Research Valparaiso, Valparaiso, Indiana
  - University of Iowa, Iowa City, Iowa
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - AMR Clinical, Lexington, Kentucky
  - Ochsner Clinic Foundation, Kenner, Louisiana
  - Ochsner Medical Center - Kenner, Kenner, Louisiana
  - Velocity Clinical Research, Metairie, Metairie, Louisiana
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - ActivMed Practices & Research, LLC, Beverly, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Michigan Center of Medical Research (MICHMER), Farmington Hills, Michigan
  - Ascension St. John Hospital Vaccine Research Unit, Grosse Pointe Woods, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Saint Louis University, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Skyline Medical Center, PC/CCT Research, Elkhorn, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Wr-Crcn, Llc., Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - ActivMed Practices and Research, LLC., Portsmouth, New Hampshire
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Velocity Clinical Research, Binghamton, Binghamton, New York
  - Drug Trials America, Hartsdale, New York
  - Corning Center for Clinical Research, Horseheads, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - CHEAR Center LLC, The Bronx, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - Atrium Health - Strive Vaccine Research Clinic, Charlotte, North Carolina
  - Tryon Medical Partners, PLLC, Charlotte, North Carolina
  - Accellacare - Charlotte, Charlotte, North Carolina
  - Sensenbrenner Primary Care Research Office, Charlotte, North Carolina
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Velocity Clinical Research, Cincinnati, Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Springdale, Cincinnati, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Tekton Research, LLC., Edmond, Oklahoma
  - Tekton Research, Inc, Yukon, Oklahoma
  - The Corvallis Clinic, PC, Corvallis, Oregon
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Summit Headlands, LLC, Portland, Oregon
  - Kaiser Permanente Northwest Center for Health Research, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Penn Prevention Unit, Philadelphia, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - AMR Clinical, Knoxville, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Innovo Research - Austin Regional Clinic, Austin, Texas
  - Tekton Research, LLC., Austin, Texas
  - Tekton Research, LLC., Beaumont, Texas
  - Javara - Privia Medical Group Gulf Coast - The Woodlands HWH, Conroe, Texas
  - North Texas Infectious Diseases Consultants, P.A, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Family Care, Fort Worth, Texas
  - Allure Health at Mt. Olympus Medical Research, Friendswood, Texas
  - Hany H. Ahmed, MD, Houston, Texas
  - Helios Clinical Research - HOU, Houston, Texas
  - HG Pediatrics, Houston, Texas
  - Trio Clinical Trials, LLC, Houston, Texas
  - Van Tran Family Practice, Houston, Texas
  - Ventavia Research Group, LLC, Houston, Texas
  - Centex Studies, Houston, Texas
  - DM Clinical Research - Cy Fair, Houston, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - DM Clinical Research - Humble, Humble, Texas
  - DM Clinical Research, Martin Diagnostic Clinic, Humble, Texas
  - Milton Haber, M.D., Laredo, Texas
  - Milton Haber, MD, Laredo, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Sun Research Institute, San Antonio, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Sugar Land, Texas
  - Javara Inc., Sugar Land, Texas
  - Mt Olympus Medical Research, Sugar Land, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic Draper, Draper, Utah
  - Tanner Clinic, Layton, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Centricity Research Suffolk Primary Care, Suffolk, Virginia
  - Virginia Gastroenterology Clinical Research, Suffolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Sound Medical Research, Port Orchard, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - MultiCare Medical Group, Tacoma, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
  - Research Building, Wenatchee, Washington
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Argentina (8):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, CABA, Buenos Aires
  - Fundación Respirar, CABA, Buenos Aires
  - Clinica Privada Instituto Medico Platense S.A., La Plata, Buenos Aires
  - Instituto De Investigaciones Clínicas Mar Del Plata, Mar del Plata, Buenos Aires
  - Clinica Mayo de Urgencias Medicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Hospital de Clinicas Presidente Nicolas Avellaneda, San Miguel de Tucumán, Tucumán Province
  - Clinica Privada del Sol S.A., Córdoba
  - IMAC - Instituto Medico de Alta Complejidad, Salta
- Canada (15):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - University Of Alberta Hospital, Edmonton, Alberta
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Dawson Clinical Research Inc, Guelph, Ontario
  - Premier Clinical Trial Network, Hamilton, Ontario
  - Centricity Research Toronto LMC Multispecialty, Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Centricity Research Toronto Manna Multispecialty, Toronto, Ontario
  - Centricity Research Mirabel Multispecialty, Mirabel, Quebec
  - Clinique de Médecine Urbaine du Quartier Latin, Montreal, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Diex Recherche Inc. Division Victoriaville, Victoriaville, Quebec
  - Diex Recherche Quebec, Québec
  - Centre de Recherche Saint-Louis inc., Québec
- Finland (13):
  - Espoo Vaccine Research Clinic, Espoo
  - FVR, Etelä-Helsingin rokotetutkimusklinikka, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Järvenpää Vaccine Research Clinic, Jarvenpaa
  - Terveystalo Jyväskylä, Jyväskylä
  - Kokkola Vaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Terveystalo Tampere, Tampere
  - Terveystalo Turku Pulssi, Turku
  - Turku Vaccine Research Clinic, Turku
- Japan (18):
  - Tenjin General Clinic, Fukuoka, Fukuoka
  - Seishinkai Inoue Hospital, Itoshima, Fukuoka
  - Sasaki Clinic, Amagasaki, Hyōgo
  - Motomachi Takatsuka Naika Clinic, Yokohama, Kanagawa
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Sugiura Clinic, Kawaguchi, Saitama
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Tokyo Eki Center Building Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Medical Corp. Seikoukai New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Hillside Clinic Jingumae, Shibuya-ku, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Oda Clinic, Shinjuku-ku, Tokyo
  - Souseikai Sumida Hospital, Sumida-ku, Tokyo
  - Sekino Hospital, Toshima-ku, Tokyo
  - SOUSEIKAI PS Clinic, Fukuoka
  - AMC Nishiumeda Clinic, Osaka
- Netherlands (11):
  - Meander Medisch Centrum, Amersfoort
  - PoliDirect Amsterdam West, Amsterdam
  - Huisartsencentrum Parklaan, Eindhoven
  - Huisartsenpraktijk Radesingel, Groningen
  - Gezondheidscentrum Leonardus, Helmond
  - Spaarne Gasthuis, Hoofddorp
  - PoliDirect Nieuwegein, Nieuwegein
  - Franciscus Gasthuis & Vlietland, location Gasthuis, Rotterdam
  - Huisartsen Soest, Soest
  - UMC Utrecht, Utrecht
  - Julius Clinical Breda, Zeist
- South Africa (21):
  - Josha Research, Bloemfontein, Free State
  - Welkom Clinical Trial Centre (MERC WELKOM), Welkom, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - MERCLINCO (Pty) Ltd - Kempton, Kempton Park, Gauteng
  - Dr A Jacovides & Partners Inc., Midrand, Gauteng
  - Newtown Clinical Research Centre (PTY) LTD, Newtown, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - About Allergy, Pretoria, Gauteng
  - Into Research, Pretoria, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Synexus SA- Watermeyer Clinical Research Center, Pretoria, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - Wits Vaccines & Infectious Diseases Analytics, Soweto, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - MERC Research (Pty) Ltd - Middelburg, Middelburg, Mpumalanga
  - Synexus - Helderberg Clinical Research Centre - Somerset West, Cape Town, Western Cape
  - TREAD Research, Cape Town, Western Cape
  - Be Part Yoluntu Centre, Paarl, Western Cape
  - Helderberg Clinical Trials Centre, Somerset West, Western Cape
  - Emmed Research, Pretoria
  - Botho Ke Bontle Health Services, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Walsh EE, Eiras D, Woodside J, Jiang Q, Patton M, Marc GP, Llapur C, Ramet M, Fukushima Y, Hussen N, Cardona J, Mikati T, Zareba A, Ilangovan K, Lino MM, Kalinina EV, Swanson KA, Gurtman A, Munjal I. Efficacy, Immunogenicity, and Safety of the Bivalent RSV Prefusion F (RSVpreF) Vaccine in Older Adults Over 2 RSV Seasons. Clin Infect Dis. 2025 Feb 10:ciaf061. doi: 10.1093/cid/ciaf061. Online ahead of print. PMID 39928572
- [Derived] Walsh EE, Perez Marc G, Zareba AM, Falsey AR, Jiang Q, Patton M, Polack FP, Llapur C, Doreski PA, Ilangovan K, Ramet M, Fukushima Y, Hussen N, Bont LJ, Cardona J, DeHaan E, Castillo Villa G, Ingilizova M, Eiras D, Mikati T, Shah RN, Schneider K, Cooper D, Koury K, Lino MM, Anderson AS, Jansen KU, Swanson KA, Gurtman A, Gruber WC, Schmoele-Thoma B; RENOIR Clinical Trial Group. Efficacy and Safety of a Bivalent RSV Prefusion F Vaccine in Older Adults. N Engl J Med. 2023 Apr 20;388(16):1465-1477. doi: 10.1056/NEJMoa2213836. Epub 2023 Apr 5. PMID 37018468
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671013